CLINICAL TRIAL: NCT06543121
Title: Validation And Turkish Cross-Cultural Adaptation of Stroke Knowledge Test
Status: Completed | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Furkan Çakır, Principal Investigator, Istanbul Bilgi University
Other Study IDs: IstanbulBUFC6
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Hypertension
Keywords: Stroke Knowledge Test; stroke education; validity; reliability
MeSH Terms: conditions — Stroke; Hypertension | interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients
  Interventions: Other: Translating the Stroke Knowledge Test into Turkish and Related Processes; Other: Validity; Other: Internal consistency and Reliability
- Hypertension patients
  Interventions: Other: Translating the Stroke Knowledge Test into Turkish and Related Processes; Other: Validity; Other: Internal consistency and Reliability

INTERVENTIONS:
Other: Translating the Stroke Knowledge Test into Turkish and Related Processes — The first step is the translation from the original language to the other language. The ideal target in the translation phase is to use people who are familiar with the structure of the original language and who are familiar with the language. Two forward translation and one reverse translation methods will be applied after obtaining the written permission of the authors. After the completion of this phase, the terminological differences arising from the translators in the translation process from the original language to Turkish will be collected and discussed on the questions. The cultural adaptation study will be terminated by determining the equivalence between the Turkish version of the test and the English original. The final version of the questionnaire and the necessary changes will be arranged specific to the investigator's society and the authors of the original questionnaire will be consulted and the questionnaire will be finalized.
Other: Validity — Content validity will be calculated with the Content Validity Index, which is a result of 10 expert opinions in terms of clarity, difficulty, and suitability of the Turkish version of the Stroke Knowledge Test. For face validity, the final version of the form will be provided with opinions from 3 stroke patients.
Other: Internal consistency and Reliability — The internal consistency of the items will be tested with Cronbach alpha. Test-retest reliability will be tested with intraclass correlation coefficient.

SUMMARY:
Cerebrovascular diseases are the leading cause of disability, work loss, and quality of life reduction, the third leading cause of death globally, and significantly impact hospital admissions and expenses. This prevalence rises with an aging population and comorbidities. Recognizing stroke symptoms quickly is crucial for timely treatment. Miscommunication or misunderstanding among hypertensive patients, who are at the highest risk for stroke, increases stroke risk and complications. Educating the public about stroke symptoms and responses is essential for prevention. Therefore, a valid and reliable tool to assess hypertensive patients' stroke knowledge is important for improving long-term outcomes. This research aims to adapt the Stroke Knowledge Test into Turkish and evaluate its validity and reliability in hypertensive patients.

DETAILED DESCRIPTION:
Cerebrovascular diseases are the group of diseases that cause the most disability and loss of work, affect the quality of life the most and are the third leading cause of death in the world, and also have a significant place in hospital admissions and expenses. This rate increases with the aging population and comorbidities. The recognition of stroke symptoms by the society is the most important factor in patients reaching treatment opportunities without wasting time.

It is known that failure to provide accurate information to hypertensive patients, who are the highest risk group for stroke, or the patient's failure to understand stroke is associated with a higher risk of stroke and complications. These findings indicate that it is important to provide information to the public about how they behave when they encounter symptoms related to stroke and related conditions. Measuring stroke knowledge and risk factors in hypertensive and potential stroke patients can serve as a healthcare provider who informs the society to adopt stroke prevention behaviors.

Therefore, a valid and reliable assessment tool is of great importance in determining whether hypertensive patients have sufficient knowledge about stroke and improving the long-term clinical outcomes of stroke.

This research aims to perform the cross-cultural adaptation of the Stroke Knowledge Test into Turkish and to examine the validity and reliability of the assessment tool in hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Native Turkish and literate
* Diagnosed with hypertension / history of ischemic or hemorrhagic stroke and
* Patients who signed the voluntary consent form will be included.

Exclusion Criteria:

* Participants who are illiterate and
* Participants who have mental problems that may prevent them from answering the test will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with stroke or hypertension
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Stroke Knowledge Test | T0 and T1 (Baseline and after 1 week after)
  It consists of 20 questions. Each question has a single correct answer from one of the 5 options, "I don't know"; this increases the validity of the questionnaire by preventing the participant from guessing the correct answer. One point is given for each correct answer, no points are given for wrong or "I don't know" answers. The scores of the 20 questions are added up and a higher score indicates a higher stroke knowledge. The content of the original scale was selected based on a review of the literature as well as the clinical experience of the original authors regarding factors determined to be important for the education of stroke patients. The items in the original scale cover the signs, symptoms and risk factors of stroke as well as factors related to the prevention, prevalence, treatment and recovery of stroke. The internal consistency α value of the original SKT is 0.65 and the test-retest reliability r value is 0.82.
Nottingham Health Profile | Baseline
  Divergent validity will be assessed with the Nottingham Health Profile. It is a general health status measurement that measures patients' quality of life in physical, emotional and social areas. The Nottingham Health Profile consists of a total of 38 items, including physical mobility (8 items), pain (8 items), sleep (5 items), emotional reactions (9 items), social isolation (5 items) and energy level (3 items). Each item is answered as "yes" or "no". A score of 0 is given for a "no" answer and a score of 1 is given for a "yes" answer. The sum of the positive answers in each section is divided by the total number of statements in that section and the result is multiplied by 100 to obtain possible results between 0 and 100. A score close to 100 indicates a low quality of life.The internal consistency α value of the measurement tool is 0.87 and the test-retest reliability r value is 0.88.

CONTACTS AND LOCATIONS:
Overall Officials: Mine Gulden Polat, Prof, Principal Investigator — Marmara University
Locations (1):
- İstanbul BilgiUniversity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided